CLINICAL TRIAL: NCT02336178
Title: An Open-label, Single-arm, Post-authorization Pragmatic Clinical Trial On The Safety And Efficacy Of Benefix (Nonacog Alfa, Recombinant Factor Ix) In Subjects With Hemophilia B In Usual Care Settings In China
Brief Title: Safety and Efficacy of Benefix in Patients With Hemophilia B in Usual Care Settings in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B1821052; 2016-000765-22 (EudraCT Number)
Record Dates: First submitted 2014-12-16; First posted 2015-01-12 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: HEMOPHILIA B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Benefix (Experimental): This is a single arm study. Subjects will be treated with Benefix by the investigator according to usual care in China and in accord with the China BeneFIX Package Insert.
  Interventions: Drug: Benefix

INTERVENTIONS:
Drug: Benefix — Subjects will be treated by the investigator according to usual care in China and in accord with the China BeneFIX Package Insert.
  The treatment duration is approximately 6 months (±7 days) or approximately 50 Exposure Days (EDs) (±5 EDs) (see protocol definition on EDs) whichever occurs first.

SUMMARY:
The purpose of this post-approval study is to evaluate the safety and efficacy of Benefix in subjects with hemophilia B in usual care settings in China.

DETAILED DESCRIPTION:
The purpose of this post-approval study is to provide supplementary information relating to the use of BeneFIX in Chinese subjects with hemophilia B, especially on the safety and efficacy in different populations of Chinese hemophilia B patients, in particular in pediatric patients <6 years of age, pediatric patients ≥6 to ≤12 years of age, Previously Untreated Patients (PUPs) , subjects receiving prophylaxis treatment after enrollment in the study, and severe patients (FIX activity <1%).

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects with hemophilia B.
* Subjects/parents/legal representatives must be able to comply with study procedures (informed consent/assent process, clinical visits, reporting of infusion and bleed data, reporting of adverse events, etc)

Exclusion Criteria:

* Presence of any other bleeding disorder in addition to hemophilia B. Subjects with a past history of, or current factor IX inhibitor. For laboratory-based assessments, any Bethesda inhibitor titer greater than the laboratory's normal range or ≥0.6 Bethesda Unit (BU)/mL.
* Subjects with known hypersensitivity to the active substance or to any of the excipients of BeneFIX.
* Subjects with a known hypersensitivity to Chinese Hamster Ovary cell proteins.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- China (16):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Centre-South University, Changsha, Hunan
  - Department of Hematology,The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Hematology,The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Department of Hematology,Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Blood Center of Shandong Province, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai JiaoTong University School of Medicine/Hematology Department, Shanghai, Shanghai Municipality
  - Shanxi Medical University Second Hospital, Taiyuan, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Blood Diseases Hospital, Chinese Academy of Medical Science (Institute of Hematology), Tianjin, Tianjin Municipality
  - Department of Hematology,The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hematology Department,Beijing Children's Hospital, Capital Medical University, Beijing
  - Children's Hospital of Chongqing Medical University, Chongqing

REFERENCES:
- [Derived] Yang R, Wu R, Sun J, Sun F, Rupon J, Huard F, Korth-Bradley JM, Xu L, Luo B, Liu YC, Rendo P. First open-label, single-arm, prospective study of real-world use of FIX replacement therapy in a predominantly pediatric hemophilia B population in China. Medicine (Baltimore). 2021 May 28;100(21):e26077. doi: 10.1097/MD.0000000000026077. PMID 34032739
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1821052&StudyName=Safety%20and%20Efficacy%20of%20Benefix%20%28nonacog%20Alfa%2C%20Recombinant%20%20Factor%20Ix%29%20in%20Patients%20with%20Hemophilia%20B%20in%20Usual%20Care%20Settings%20in%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 70 participants.
Groups:
- BeneFIX: Participants received intravenous (IV) infusions of BeneFIX for on-demand or prophylaxis treatment at a dose and frequency prescribed by the participant's treating physician in accordance with the China BeneFIX Package Insert for 6 months (±7 days) or 50 Exposure Days (EDs) (±5 EDs), whichever occurred first.
Period: Overall Study
Arm/Group | BeneFIX
Started | 70
Completed | 66
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all enrolled participants who received the study drug.
Arm/Group | BeneFIX
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Factor IX Inhibitor
Description: Factor IX (FIX) inhibitor development was defined as any Bethesda inhibitor titer greater than the laboratory's normal range or Bethesda inhibitor titer >=0.6 Bethesda Unit (BU)/mL.
Time Frame: Up to 6 months
Population: All participants who received at least 1 dose of BeneFIX during the study. Participants in each arm were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pediatric Participants <6 Years of Age; Pediatric Participants ≥6 to ≤12 Years of Age; Previously Untreated Participants (PUPs); Severe Participants (Factor IX Activity <1%): Participants received intravenous (IV) infusions of BeneFIX for on-demand or prophylaxis treatment at a dose and frequency prescribed by the participant's treating physician in accordance with the China BeneFIX Package Insert for 6 months (±7 days) or 50 Exposure Days (EDs) (±5 EDs), whichever occurred first.
- Participants Receiving Prophylaxis Treatment: Participants received intravenous (IV) infusions of BeneFIX for on-demand or prophylaxis treatment at a dose and frequency prescribed by the participant's treating physician in accordance with the China BeneFIX Package Insert for 6 months (±7 days) or 50 Exposure Days (EDs) (±5 EDs), whichever occurred first. This reporting arm included all participants who received prophylaxis treatment after enrollment in the study.
- Overall Participants: Participants received intravenous (IV) infusions of BeneFIX for on-demand or prophylaxis treatment at a dose and frequency prescribed by the participant's treating physician in accordance with the China BeneFIX Package Insert for 6 months (±7 days) or 50 Exposure Days (EDs) (±5 EDs), whichever occurred first. This reporting arm included all participants who received at least 1 dose of BeneFIX during the study.
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 30 | 31 | 11 | 57 | 36 | 70
percentage of participants | 3.3 [0.1 to 17.2] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 28.5] | 1.8 [0.0 to 9.4] | 0.0 [0.0 to 9.7] | 1.4 [0.0 to 7.7]

2. Primary Outcome: Number of Participants With Allergic Reactions
Description: FIX product allergy was defined as a hypersensitivity reaction to a FIX product with symptoms such as hives, urticaria, tightness of chest, wheezing, hypotension, and anaphylaxis based on investigator's judgments.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 30 | 31 | 11 | 57 | 36 | 70
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Thrombotic Events
Description: Thrombotic event was defined as any event associated with formation of a blood clot including catheter-associated thrombi and thrombotic complications.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 30 | 31 | 11 | 57 | 36 | 70
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causality with the treatment or usage. A serious adverse event (SAE) was any untoward occurrence at any dose that resulted in death; was life threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both serious and non-serious AEs. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study drug.
Time Frame: Up to 7 months (28 calendar days after end of 6-month or 50-exposure day study treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 30 | 31 | 11 | 57 | 36 | 70
participants
  AEs | 28 | 26 | 10 | 46 | 30 | 62
  SAEs | 2 | 0 | 0 | 2 | 0 | 2

5. Secondary Outcome: Annualized Bleeding Rates (ABRs) in Participants Receiving Prophylaxis Treatment With BeneFIX During Their Prophylaxis Period
Description: For prophylaxis period, annualized bleeding rate (ABR) was derived for each participant by the following formula: ABR = number of bleeds in prophylaxis period / (number of days in prophylaxis period/365.25). A prophylaxis period was defined as time from first prophylaxis infusion through 6 calendar days after the day of last prophylaxis infusion, or the day of study conclusion visit, whichever was earlier. A break in the prophylaxis period was any period of 28 days or longer in which no prophylaxis infusions were given. For a prophylaxis regimen to have been qualified to have ABR calculated, the sum of its periods needed to be >=14 days.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants who participated in at least 1 day of a prophylaxis period (ie, had at least 1 prophylaxis dose). Participants in each arm were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: episodes/year
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 27 | 28 | 7 | 57 | 29 | 57
episodes/year | 5.9 (9.46) | 7.5 (8.97) | 0.3 (0.72) | 6.5 (9.06) | 5.5 (7.94) | 6.5 (9.06)

6. Secondary Outcome: Number of Spontaneous/Non-traumatic Breakthrough Bleeds Within 48 Hours of a Prophylaxis Dose of BeneFIX
Description: The prophylaxis infusion time, bleed start time and bleed type (etiology) were used to determine the number of spontaneous, non-traumatic breakthrough bleeds that occurred <=48 hours after a prophylaxis infusion. If there was more than 1 bleed location (eg, ankle and joint) with identical bleed start date and time, it was treated as 1 bleed occurrence.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants with any spontaneous/non-traumatic breakthrough bleeds within 48 hours of a prophylaxis dose. Participants in each arm were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: breakthrough bleeds
Units Other Than Participants: Prophylaxis Infusions with Bleeds
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 4 | 7 | 0 | 11 | 7 | 11
Number analyzed (Prophylaxis Infusions with Bleeds) | 5 | 18 | 0 | 23 | 18 | 23
breakthrough bleeds | 1.3 (0.50) | 2.6 (2.30) |  | 2.1 (1.92) | 2.6 (2.30) | 2.1 (1.92)

7. Secondary Outcome: Annualized Bleeding Rates (ABRs) in Participants Receiving On-demand Treatment With BeneFIX During Their On-demand Period
Description: For on-demand period, the annualized bleeding rate (ABR) was derived for each participant by the following formula: ABR = number of bleeds in on-demand period / (number of days in on-demand period/365.25). The on-demand period was defined as the entire time of enrollment in the study (ie, from the date of the enrollment visit through the day before the Final/Early Termination visit) except time in any prophylaxis period. The breaks in the prophylaxis period were considered on-demand periods. For an on-demand regimen to have been qualified to have ABR calculated, the sum of its periods needed to be >= 14 days.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants who received on-demand treatment during on-demand period. Participants in each arm were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: episodes/year
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 5 | 6 | 4 | 10 | 18
episodes/year | 14.8 (15.59) | 28.2 (26.16) | 6.2 (2.40) | 29.3 (25.95) | 26.3 (23.08)

8. Secondary Outcome: Number of Infusions Resulted in the Following Response to On-demand Treatment of Bleeds: Excellent, Good, Moderate, no Response
Description: Response was assessed using 4-point On-Demand Hemostasis Efficacy Rating Scale. Excellent means definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with no additional infusion administered; good means definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with at least one additional infusion administered for complete resolution of the bleeding episode, or definite pain relief and/or improvement in signs of bleeding starting after 8 hours following the infusion, with no additional infusion administered; moderate means probable or slight improvement starting after 8 hours following the infusion, with at least one additional infusion administered for complete resolution of the bleeding episode; no response means no improvement between infusions or during the 24 hour interval following an infusion, or condition worsens. Both first infusions and follow-up infusions were included.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants who had a bleed during the study for which on-demand treatment with BeneFIX was administered. Participants in each arm were not mutually exclusive.
Measure: Number; unit: infusions
Units Other Than Participants: Infusions
Groups:
- Participants Receiving Prophylaxis Treatment: Participants received prophylaxis treatment with BeneFIX according to usual care in China and in accord with the China BeneFIX Package Insert. The treatment duration was 6 months (±7 days) or 50 Exposure Days (±5 EDs) whichever occurred first. On-demand treatment was given as needed.
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 18 | 20 | 5 | 32 | 24 | 46
Number analyzed (Infusions) | 164 | 211 | 18 | 249 | 302 | 520
infusions
  Excellent | 77 | 94 | 9 | 133 | 122 | 254
  Good | 60 | 91 | 9 | 96 | 145 | 204
  Moderate | 22 | 23 | 0 | 19 | 33 | 54
  No response | 5 | 3 | 0 | 1 | 2 | 8

9. Secondary Outcome: Number of BeneFIX Infusions to Treat Each New Bleed
Description: The number of BeneFIX infusions administered to treat each new bleed was calculated by adding the on-demand initial treatment and any on-demand follow-up treatments for the same bleed. If there was more than one bleed location (eg, ankle and joint) with identical bleed start date and time, it was treated as one bleed occurrence.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: infusions
Units Other Than Participants: Bleeds
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 18 | 20 | 5 | 32 | 24 | 46
Number analyzed (Bleeds) | 96 | 137 | 16 | 162 | 198 | 353
infusions | 1.7 (1.72) | 1.5 (2.03) | 1.1 (0.34) | 1.5 (1.23) | 1.5 (2.01) | 1.5 (1.71)

10. Secondary Outcome: Average Infusion Dose and Total Factor IX Consumption in On-demand Setting
Description: The total amount (international units [IU]) infused for each BeneFIX infusion was summed to calculate the total factor IX consumption for each participant. The average infusion dose for each participant was calculated as his total factor IX consumption (in IU) divided by the number of infusions administered.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 18 | 20 | 5 | 32 | 24 | 46
IU
  Total FIX consumption | 4277.8 (4659.47) | 6550.0 (6540.66) | 1770.0 (1173.46) | 4418.8 (3449.75) | 11672.9 (16304.85) | 9826.1 (14816.34)
  Average infusion dose | 451.1 (161.44) | 658.5 (370.35) | 518.6 (295.70) | 607.7 (309.34) | 803.8 (549.75) | 731.6 (498.58)

11. Secondary Outcome: Average Infusion Dose and Total Factor IX Consumption in Prophylaxis Setting
Description: as for outcome 10
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants who received at least 1 dose of prophylaxis BeneFIX treatment during the study. Participants in each arm were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 27 | 28 | 7 | 57 | 29 | 57
IU
  Total FIX consumption | 14709.3 (8910.57) | 22102.7 (18860.51) | 13846.4 (5868.21) | 19224.1 (15424.70) | 20628.4 (19894.00) | 19224.1 (15424.70)
  Average infusion dose | 429.3 (193.52) | 623.1 (377.99) | 351.9 (194.48) | 540.1 (316.56) | 557.0 (407.05) | 540.1 (316.56)

12. Secondary Outcome: Average Infusion Dose and Total Factor IX Consumption in Recovery Setting
Description: as for outcome 10
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: All participants who received at least 1 recovery infusion with BeneFIX during the study. Participants in each arm were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 12 | 9 | 1 | 20 | 13 | 24
IU
  Total FIX consumption | 1156.3 (1341.14) | 1688.9 (1123.27) | 250.0 (NA) — Analysis population only included 1 participant, therefore, the standard deviation was not calculated. | 1378.8 (1291.66) | 1467.3 (1318.28) | 1419.8 (1192.62)
  Average infusion dose | 773.4 (371.46) | 890.7 (270.46) | 250.0 (NA) — Analysis population only included 1 participant, therefore, the standard deviation was not calculated. | 889.9 (502.77) | 962.0 (556.45) | 929.1 (475.75)

13. Secondary Outcome: Percentage of Infusions With Less Than Expected Therapeutic Effects (LETEs) in On-demand Setting
Description: Less than expected therapeutic effect (LETE) in the on-demand setting was defined as 2 successive "no response" ratings recorded after 2 successive BeneFIX drug infusions, respectively.
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of infusions
Units Other Than Participants: Bleeding Episodes
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 18 | 20 | 5 | 32 | 24 | 46
Number analyzed (Bleeding Episodes) | 96 | 137 | 16 | 162 | 198 | 353
percentage of infusions | 0 [0 to 3.8] | 0 [0 to 2.7] | 0 [0 to 20.6] | 0 [0 to 2.3] | 0 [0 to 1.8] | 0 [0 to 1.0]

14. Secondary Outcome: Percentage of Infusions With Less Than Expected Therapeutic Effects (LETEs) in Prophylaxis Setting
Description: Less than expected therapeutic effect (LETE) in the prophylaxis setting was defined as occurrence of any spontaneous bleed within 48 hours after a regularly scheduled prophylactic dose of BeneFIX (which was not used to treat a bleed).
Time Frame: Up to 6 months or 50 exposure days whichever occurred first
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of infusions
Units Other Than Participants: Prophylaxis Infusions
Arm/Group | Pediatric Participants <6 Years of Age | Pediatric Participants ≥6 to ≤12 Years of Age | Previously Untreated Participants (PUPs) | Participants Receiving Prophylaxis Treatment | Severe Participants (Factor IX Activity <1%) | Overall Participants
Number analyzed (Participants) | 27 | 28 | 7 | 57 | 29 | 57
Number analyzed (Prophylaxis Infusions) | 934 | 1006 | 287 | 2032 | 1069 | 2032
percentage of infusions | 0.1 [0 to 0.6] | 0.1 [0 to 0.6] | 0 [0 to 1.3] | 0.1 [0 to 0.4] | 0.2 [0.0 to 0.7] | 0.1 [0 to 0.4]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | BeneFIX
Serious Adverse Events (participants affected / at risk) | 2/70
Other Adverse Events (participants affected / at risk) | 55/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeneFIX (N=70)
Factor IX inhibition (Blood and lymphatic system disorders) | 1 (1)
Oral mucosa haematoma (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeneFIX (N=70)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Peripheral swelling (General disorders) | 6 (9)
Pyrexia (General disorders) | 11 (18)
Nasopharyngitis (Infections and infestations) | 19 (27)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Contusion (Injury, poisoning and procedural complications) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (76)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 6 (20)
Joint swelling (Musculoskeletal and connective tissue disorders) | 15 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.